CLINICAL TRIAL: NCT01811238
Title: A Multicenter, Phase IV, Interventional Study to Assess the Efficacy and Safety of TARGIN(R) (Oxycodone/Naloxone) in Korean Patients With Spinal Disorders
Brief Title: An Interventional Study to Assess the Efficacy and Safety of Oxycodone/Naloxone in Korean Patients With Spinal Disorders
Acronym: TALENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OXN12-KR-401
Record Dates: First submitted 2012-10-22; First posted 2013-03-14 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Spinal Disorders
Keywords: spinal disorders
MeSH Terms: interventions — Oxycodone; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxycodone/Naloxone (Experimental): Single-arm study
  Interventions: Drug: Oxycodone/naloxone

INTERVENTIONS:
Drug: Oxycodone/naloxone — Targin 5mg, 10mg, 20mg up to 40mg b.i.d
  Other Names: Targin

SUMMARY:
Study Objectives:

1. Primary objective

   - To assess the pain reduction after 8 weeks treatment from baseline (week 0)
2. Secondary objectives

   * To assess the pain reduction after 4 weeks treatment from baseline (week 0)
   * To assess the EQ-5D
   * To assess physician's overall satisfaction
   * To assess subject's overall satisfaction
   * To assess safety

DETAILED DESCRIPTION:
Study Design (Methodology):

This will be a multicenter, phase IV, interventional study to assess the efficacy and safety of TARGIN(R)(Oxycodone/Naloxone) in Korean patients who are dissatisfied with their current analgesic medication (WHO step II analgesics).

Upon providing written informed consent, subject will be screened in the study and assessment will be performed at that time such as safety laboratory assessments, physical examination, vital sign, medical history taking, 24 hours pain intensity score, EQ-5D, physician's overall satisfaction and subject's overall satisfaction. If patient is eligible in inclusion/exclusion criteria at the time of visit 1, the patient will receive treatment with TARGIN(R). Re-screening, study drug dose interruption is not allowed. The duration of study drug dose interruption is defined as for 1 week.

Treatment with TARGIN(R) will be started at 5/2.5mg b.i.d.,and proper titration (up titration) will be allowed at each visit or at unscheduled visit according to the investigator's decision. On-site visit or phone call will be allowed for visit 2(wk 1).The up titration will be considered by investigator's judgement as followings; (1) if the rescue medication was used more than 2 times per day, on average or (2) based on the daily average numerical rating scale

, if the numerical rating scale was changed to worsen since the previous visit, (3) Investigator's judgement by considering any titration needed situation (e.g. dose, frequency of rescue medication). Pain assessment by investigator at each visit will be used for analysis and criteria for uptitration. Daily pain diary will be used for only criteria for uptitration.

Safety laboratories will be obtained at baseline (visit 1) and study end (visit 4) in a local laboratory. The laboratory values within 4 weeks prior to baseline (visit 1) will be allowed to use at study visit 1.

The rescue medication is the IRcodon(R).

Patients will be withdrawn from the study if the following circumstance require study drug discontinuation:

* Failure of pain control (Failure of pain control will be decided by investigators judgement, e.g. there is poor pain control or lack of efficacy despite 2~3 times of titration.)
* Adjustment of the other analgesics due to Adverse event except TARGIN(R) or IRcodon(R)
* Adjustment of the other major pain management modality (e.g. surgery, non-surgical interventional therapy, etc.)
* Withdrawal of informed consent
* Pregnancy
* Any other significant risk to the patient's safety in the clinical judgement of the investigator

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 20 and <80 years of age
* Patients who have spinal disorders related pain for over 90days
* Patients who have moderate to severe pain intensity which is not controlled with weak opioids or NSAIDs: NRS ≥ 4
* Naïve patients for Oxycodone/Naloxone
* Naïve patients for strong opioid
* Patients who signed a written informed consent form

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
* Patients with known hypersensitivity to Oxycodone/Naloxone or to any of the excipients
* Patients with severe respiratory depression with hypoxia and/or hypercapnoea
* Patients with severe chronic obstructive pulmonary disease
* Patients with cor pulmonale
* Patients with severe bronchial asthma
* Patients who have been diagnosed or is suspected of having paralytic or obstructive ileus.Patients with moderate to severe hepatic impairment
* Targin(R) product contains lactose. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take
* Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels (>2.5 times the upper limit of normal, it is allowed >5 times the upper limit of normal in case of transition in liver) or an abnormal total bilirubin and/or creatinine level (s)(greater than 1.5 times the upper limit of normal), gamma glutamyl transpeptidase (GGT or GGTP) ≥ 3 times the upper limit of normal
* Patients with uncontrolled seizures
* Requiring interventional treatment for pain such as neurodestructive procedure or regional infusion
* Patients with increased intracranial pressure
* In the investigator's opinion, subjects who are receiving hypnotics or central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study medication
* Patients with myxodema, not adequately treated hypothyroidism or Addisons disease
* Patients receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine)
* Clinically significant impairment of cardiovascular, respiratory and renal function
* Major surgery within 1 month prior to screening or planned surgery
* Mainly pain originated other than spinal disorders disease
* Non-malignant patients or cancer patients who are receiving any oncology treatment that could affect the measure of pain control
* Patients with uncontrolled constipation regardless of laxative use and/or laxative type
* With a disability that may prevent the patient from completing all study requirements and in particular, interfere with 24hrs pain intensity score
* Patients known to have, or suspected of having a history of drug abuse
* Patients with history of opioid or drug dependence
* Any situation where opioids are contraindicated
* Patient who needs acute dose titration or whose pain intensity fluctuate significantly in a short period according to investigator's judgment
* Having used other investigational drugs at the time of enrollment

No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Soo Shung, Principal Investigator — Samsung Medical Center

REFERENCES:
- [Derived] Hwang CJ, Chung SS, Lee KY, Lee JH, Moon SH, Kim JH, Cho KJ, Ahn JS, Kim DS, Park YS, Park HJ. Analgesic Efficacy and Safety of Prolonged-Release Oxycodone/Naloxone in Korean Patients with Chronic Pain from Spinal Disorders. Clin Orthop Surg. 2018 Mar;10(1):33-40. doi: 10.4055/cios.2018.10.1.33. Epub 2018 Feb 27. PMID 29564045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 10 general hospitals were recruited patients from 26 Sep. 2012 to 02 Aug. 2013.
Groups:
- Oxycodone/Naloxone: Single-arm study
  Oxycodone/Naloxone: 8 weeks treatment with Oxycodone/Naloxone
Period: Overall Study
Arm/Group | Oxycodone/Naloxone
Started | 240 (First patient was recruited on 26 Sep. 2012.)
Safety Set | 220 (20 subjects excluded from the safety set due to study drug not administered.)
ITT Set | 209 (11 subjects excluded from ITT set due to no primary efficacy assessment(5) and IC/EC violation(6).)
PP Set | 120 (89 subjects excluded from PP set due to various reasons.)
Completed | 159 (159 subjects regardless PP set completed study visit.)
Not Completed | 81
Not completed — Withdrawal by Subject | 42
Not completed — Adverse Event | 25
Not completed — Protocol Violation | 4
Not completed — Lack of Efficacy | 4
Not completed — subject refused study medication | 6

BASELINE CHARACTERISTICS:
Population: Total 240 patients were enrolled. However, 20 patients were excluded due to no administeration of investigational drug during the study. The 220 is Safety set population included all subjects who had at least one dose of the study drug.
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.25 (10.42)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 86
  >=65 years | 134
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 84
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 220

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Intensity of Patient With Spinal Disorder as Measured by NRS.
Description: NRS-Pain scale assessed the severity of a subject's pain of mean pain over the past 24 hours prior to the visit on a scale of 0 (No pain) and 10 (Worst possible pain).
  Change = mean score at Week 8/ET minus mean score at Baseline.
Time Frame: Baseline, 8 week
Population: The 209 is IIT set population. ITT set included all subjects who participated in the study and had at least one dose of the study drug and had at least one primary efficacy endpoint data available.
  Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 209
scores on a scale | -1.69 (2.18)
Statistical Analysis 1: Comparison: Oxycodone/Naloxone; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; The primary endpoint will be the actual reduction rate of pain intensity (0 -10) score at 8 weeks. It will be analyzed by using paired t-test; Mean Difference (Final Values) = -1.69, Standard Deviation 2.18

2. Secondary Outcome: The Change in Quality of Life (EQ-5D) at Week 8 of Treatment With the Study Drug From Baseline
Description: EQ-5D to measure of health related quality of life should be answered as one of 3 levels about current condition for 5 dimensions and was calculated total average by giving a weighting on 3 level of answers (EQ-5D levels into 'no problems' (level 1) and 'problems' (level 2 and 3)).
  Table of scores by each level for EQ-5D items: mobility(level 1=0, level2=0.069,level 3=0.314), self care(level 1=0, level2=0.104,level 3=0.214), usual activities(level 1=0, level2=0.036,level 3=0.094), pain/discomfort (level 1=0, level2=0.,level 3=0.386) and anxiety/depression(level 1=0, level2=0.071,level 3=0.2)
  *EQ-5D Total = 1 - 0.081 - (the score of the each level) - 0.269 (if at least one of level 3 presents)
  EQ-5D total score could be 0.919 in maximum and -0.594 in minimum if case all index indicates the level 3. So, if EQ-5D total score closed by "1" means that the healthy condition and high quality of life.
Time Frame: Baseline, 8 week
Population: ITT set included all subjects who participated in the study and had at least one dose of the study drug and had at least one primary efficacy endpoint data available.Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 209
scores on a scale | 0.15 (0.37)
Statistical Analysis 1: Comparison: Oxycodone/Naloxone; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; The change(difference) in EQ-5D score at Week 8 from baseline was analyzed by using paired t-test; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0 to 1.12], Standard Deviation 0.37

3. Secondary Outcome: Clinical Global Impression of Change(CGIC)
Description: The number of patients who choose the best opinion of overall satisfaction among Clinical Global Impression of Change Scale(CGIC) among 7 point scale. Missing data was imputed by LOCF.
  Very much improved much improved minimally improved no change minimally worse much worse very much worse
Time Frame: Baseline, 8 week
Population: ITT Population. Below results : Visit 4(8week)(LOCF): n(%)
Measure: Number; unit: participants
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 209
participants
  Very much improved | 20
  Much improved | 49
  Minimally improved | 70
  No change | 57
  Minimally worse | 6
  much worse | 5
  Very much worse | 2

4. Secondary Outcome: Change of Pain Intensity in Patient With Spinal Disorder at Week 4 of Treatment With the Study Drug From Baseline
Description: NRS-Pain scale assessed the severity of a subject's pain of mean pain over the past 24 hours prior to the visit on a scale of 0 (No pain) and 10 (Worst possible pain).
  Change = mean score at Week 4/ET minus mean score at Baseline.
Time Frame: Baseline, 4 week
Population: IIT set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 209
units on a scale | -1.36 (2.04)

5. Secondary Outcome: Change From Baseline in Health-related Quality of Life Assessed by EuroQol Visual Analog Scale (EQ-5D VAS)
Description: The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' (score = 100) and 'Worst imaginable health state' (score = 0). Higher points were positive results and positive points of difference gap means improvement results.
Time Frame: Baseline, 8 weeks
Population: ITT set, Missing values were imputed by LOCF. Difference (Visti 4(8w)-Baseline)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 209
scores on a scale | 10.57 (22.11)

6. Secondary Outcome: Patient Global Impression of Change(PGIC)
Description: Number of participants with categorical change in overall satisfaction. PGIC: a participant-rated instrument assessing change in participant's overall satisfaction from baseline, on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline, 8week
Population: IIT set, Missing values were imputed by LOCF.
Measure: Number; unit: participants
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 209
participants
  Very much improved | 16
  Much improved | 49
  Minimally improved | 69
  No change | 60
  Minimally worse | 6
  Much worse | 6
  Very much worse | 3

ADVERSE EVENTS:
Time Frame: Follow up 8 weeks
Description: In the safety set, a total of 120 AEs were reported in 77 subjects (35.0%, 77/220 subjects), regardless of causal relationship to the study drug. Of those, 95 events in 61 subjects (27.7%,61/220 subjects) were ADRs of which causal relationship to the study drug cannot be ruled out.
Arm/Group | Oxycodone/Naloxone
Serious Adverse Events (participants affected / at risk) | 3/220
Other Adverse Events (participants affected / at risk) | 77/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=220)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated with study drug
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related with investigational drug
Renal cancer (Renal and urinary disorders) | 1 (1) — Not related with investigational drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=220)
Nausea (Gastrointestinal disorders) | 21 (21)
constipation (Gastrointestinal disorders) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 14 (14)
Somnolence (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 4 (4)
Parosmia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (3)
Thirst (General disorders) | 2 (2)
Face oedema (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Nasopharyngitis (Infections and infestations) | 3 (3)
Cystitis (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No